CLINICAL TRIAL: NCT06050356
Title: A Phase 1a, Dose-finding, Open-label Trial Followed by a Phase 1b, Double-blind, Randomised, Placebo-controlled Trial to Evaluate the Safety, Reactogenicity, and Immunogenicity of the Tuberculosis Subunit Vaccine H107e/CAF®10b in Adults
Brief Title: First-in-Human Trial of the Novel Tuberculosis Vaccine Candidate, H107e/CAF®10b
Acronym: nTB-01
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Statens Serum Institut (Other)
Collaborators: Aurum Institute (Other); Bill and Melinda Gates Foundation (Other); Leiden University Medical Center (Other); South African Tuberculosis Vaccine Initiative (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: nTB-01; INV-042397 (Other Grant/Funding Number: Bill & Melinda Gates Foundation); DOH-27-102023-7355 (Registry Identifier: South African National Clinical Trials Registry)
Record Dates: First submitted 2023-09-17; First posted 2023-09-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: Prophylactic tuberculosis vaccine; First-in-human; Subunit vaccine; Adjuvant; BCG; Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Intervention Model Description: Phase 1a proceeds as sequential dosing to determine early safety signals (Arms 1, 2, 3, 4a, and 4b).
  Phase 1b proceeds as parallel assignment. Participants are randomised to one of four treatment arms (H107e/CAF®10b; H107e/CAF®10b + BCG; BCG; placebo).
Masking Description: Phase 1a is open label
  Phase 1b is double-blind, randomised, and placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Arm 1 (phase 1a) (Experimental): H107e
  Interventions: Biological: H107e
- Arm 2 (phase 1a) (Experimental): CAF®10b
  Interventions: Biological: CAF®10b
- Arm 3 (phase 1a) (Experimental): H107e/CAF®10b - low adjuvant dose
  Interventions: Biological: H107e/CAF®10b - low adjuvant dose
- Arm 4a (phase 1a) (Experimental): H107e/CAF®10b - full adjuvant dose - low dose intranasal H107e
  Interventions: Biological: H107e/CAF®10b - full adjuvant dose; Biological: Low dose intranasal H107e
- Arm 4b (phase 1a) (Experimental): H107e/CAF®10b - full adjuvant dose - full dose intranasal H107e
  Interventions: Biological: H107e/CAF®10b - full adjuvant dose; Biological: Full dose intranasal H107e
- Arm 1 (phase 1b) (Experimental): H107e/CAF®10b
  Interventions: Biological: H107e/CAF®10b; Biological: i.d. placebo; Biological: Intranasal H107e
- Arm 2 (phase 1b) (Experimental): H107e/CAF®10b + BCG
  Interventions: Biological: H107e/CAF®10b; Biological: BCG; Biological: Intranasal H107e
- Arm 3 (phase 1b) (Active Comparator): BCG
  Interventions: Biological: i.m. placebo; Biological: BCG; Biological: Intranasal H107e
- Arm 4 (phase 1b) (Placebo Comparator): Placebo
  Interventions: Biological: i.m. placebo; Biological: i.d. placebo; Biological: Intranasal H107e

INTERVENTIONS:
Biological: H107e — Participants will receive two i.m. injections of 20 µg unadjuvanted H107e on Day 1 and Day 29
  Arms: Arm 1 (phase 1a)
Biological: CAF®10b — Participants will receive two i.m. injections of CAF®10b (full adjuvant dose) on Day 1 and Day 29
  Arms: Arm 2 (phase 1a)
Biological: H107e/CAF®10b - low adjuvant dose — Participants will receive two i.m. injections of 20 µg H107e/CAF®10b (low adjuvant dose) on Day 1 and Day 29
  Arms: Arm 3 (phase 1a)
Biological: H107e/CAF®10b - full adjuvant dose — Participants will receive two i.m. injections of 20 µg H107e/CAF®10b (full adjuvant dose) on Day 1 and Day 29
  Arms: Arm 4a (phase 1a); Arm 4b (phase 1a)
Biological: Low dose intranasal H107e — Participants will receive one i.n. administration of 15 µg H107e (low dose intranasal H107e) on Day 85
  Arms: Arm 4a (phase 1a)
Biological: Full dose intranasal H107e — Participants will receive one i.n. administration of 30 µg H107e (full dose intranasal H107e) on Day 85
  Arms: Arm 4b (phase 1a)
Biological: H107e/CAF®10b — Participants will receive two i.m. injections of 20 µg H107e/CAF®10b (full adjuvant dose) on Day 1 and Day 29
  Arms: Arm 1 (phase 1b); Arm 2 (phase 1b)
Biological: i.m. placebo — Participants will receive two i.m. injections of placebo on Day 1 and Day 29
  Arms: Arm 3 (phase 1b); Arm 4 (phase 1b)
Biological: BCG — Participants will receive one i.d. injection of BCG on Day 1
  Arms: Arm 2 (phase 1b); Arm 3 (phase 1b)
Biological: i.d. placebo — Participants will receive one i.d. injection of placebo on Day 1
  Arms: Arm 1 (phase 1b); Arm 4 (phase 1b)
Biological: Intranasal H107e — Participants will receive one i.n. administration of 30 µg H107e (full dose intranasal H107e) on Day 211
  Arms: Arm 1 (phase 1b); Arm 2 (phase 1b); Arm 3 (phase 1b); Arm 4 (phase 1b)

SUMMARY:
Tuberculosis (TB) is an infection caused by bacteria passed from one person to another through the air when an infected person for instance coughs, speaks, or sneezes. This study tests the safety and vaccine-induced immune response of a new preventive TB vaccine called H107e/CAF®10b. H107e is a copy of protein parts from the bacterium causing tuberculosis, Mycobacterium tuberculosis, which are also called antigens. CAF®10b is an adjuvant which helps the body discover the antigen. The adjuvant and antigen are mixed together to formulate the final vaccine. The final formulated vaccine enhances the immune system's response against the antigen.

This is a first-in-human study, meaning this vaccine is being given to people for the first time. The primary objective is to evaluate the safety of the vaccine and its components; however, the study will also evaluate the specific immune responses generated by the new vaccine. The study is divided into two parts, phase 1a and phase 1b. Phase 1a investigates unadjuvanted H107e, CAF®10b adjuvant, H107e/CAF®10b vaccine (low adjuvant dose), and H107e/CAF®10b vaccine (full adjuvant dose). The trial products are administered twice intramuscularly. H107e is also administered intranasally in one of the groups on Day 85. Phase 1b investigates H107e/CAF®10b, H107e/CAF®10b+Bacillus Calmette-Guérin (BCG), BCG, and placebo. A placebo is a look-alike substance that contains no active drug. All groups in phase 1b receive H107e intranasally on Day 211.

A preventive TB vaccine such as H107e/CAF®10b should be able to introduce the body's immune system to antigens from Mycobacterium tuberculosis. This will result in memory in the immune system, meaning that when a person gets infected with Mycobacterium tuberculosis, the immune system will recognise and target the bacteria to prevent disease, thereby avoiding the need for antibiotic treatment and/or other treatments and their side effects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged ≥18 years and ≤ 45 years of age on the day of the screening visit
* Completed the written informed consent process
* Confirmed HIV-negative at screening
* Confirmed Xpert MTB/RIF Ultra-negative at screening
* Laboratory values within the indicated ranges obtained at screening:

  * Absolute neutrophil count (ANC) ≥800 cells/mm3
  * Haemoglobin ≥ 11 g/dL for females and >10.5 g/dL for males
  * Platelet count ≥ 100,000/mm3
  * Serum creatinine ≤ 1.5 X upper limit of normal (ULN)
  * AST (SGOT), ALT (SGPT), and alkaline phosphatase, ≤ 2.5 X ULN
  * Total bilirubin ≤ 2 X ULN)
* Agrees to refrain from blood donation during the course of the trial
* Women of child-bearing potential must use a highly effective form of birth control (confirmed by the investigator) throughout the trial

  * A highly effective method of birth control is defined as hormonal contraceptives (oral, injection, transdermal patch, or implant), bilateral tubal occlusion or intrauterine device. The participants must have used the contraceptive method continuously for at least 21 days prior to the pregnancy test at baseline (Day 1)
  * A female is defined as not being of child-bearing potential if she is postmenopausal (aged 50 and above with at least 12 months with no menses without an alternative medical cause prior to screening. If less than 50 years old, then confirmatory Follicular stimulating hormone testing is required)
  * A female is defined as not being of child-bearing potential if she is surgically sterile (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy). Written evidence of surgical sterility would be optimal
* Agrees to give access to medical records for trial related purposes
* Agrees to stay in contact with the trial site for the duration of the trial, provide updated contact information as necessary and has no current plans to move from the area for the duration of the trial

Exclusion Criteria:

* Previous diagnosis or current diagnosis of TB, including suspected subclinical TB
* Reported current household contact with TB. Note: Daily caregivers to TB infected persons will be considered as household contacts
* History of or ongoing severe disease that in the opinion of the investigator might affect the safety of the participant or the immunogenicity of the trial product
* Insulin-dependent diabetes
* History of allergic disease or reactions likely to be exacerbated by any component of the trial product
* History of chronic allergic rhinitis likely to interfere with the assessment of the mucosal recall
* History of frequent or severe epistaxis
* History or laboratory evidence of primary and/or acquired immunodeficiency, autoimmune disease, or immunosuppression
* History of a malignant condition (e.g. lymphoma, leukaemia, Hodgkin's disease or other tumours of the reticuloendothelial system)
* History of chronic hepatitis
* Has a body mass index ≤18 or ≥35 at screening (weight [kg] / (height [m] * height [m]))
* Abnormal chest X-ray at screening
* Receipt or planned receipt of any other investigational TB vaccine
* Receipt or planned receipt of any other investigational drug
* Receipt of emergency use authorised/emergency use listed [EUA/EUL] vaccines or licensed live attenuated vaccines (e.g., measles, mumps, and rubella [MMR], oral polio vaccine [OPV], varicella, yellow fever, live attenuated influenza vaccine, live attenuated COVID-19 vaccine) within 30 days prior to screening
* Receipt of any EUA/EUL or licensed vaccines that are not live attenuated vaccines (e.g., tetanus, pneumococcal, Hepatitis A or B, not live attenuated COVID-19 vaccine) within 14 days prior to screening
* Receipt of anticoagulant therapy, including daily acetylsalicylic acid product. NOTE: Intermittent symptomatic use is permitted
* Receipt of treatment likely to modify the immune response (e.g. blood products, immunoglobulins) within 42 days before screening
* Receipt of immunosuppressive medications, including radiotherapy, nasal corticosteroids and inhaled corticosteroids. NOTE: Use of the following is permitted:

  * Topical corticosteroids for mild, uncomplicated dermatologic conditions except if administered on the site of injection of trial products
  * A single course of oral/parenteral prednisone or equivalent at doses <60 mg/day and for <11 days with completion at least 30 days prior to screening
* Female participants: if lactating/nursing, or pregnant as per positive pregnancy test
* Not suitable for inclusion in the opinion of the investigator

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with solicited injection site reactions recorded up to seven days after each i.m. vaccination (phase 1a) | Up to Day 8 (7 days after first dose) and Day 29 up to Day 36 (7 days after second dose)
Percentage of participants with solicited systemic reactions recorded up to seven days after each i.m. vaccination (phase 1a) | Up to Day 8 (7 days after first dose) and Day 29 up to Day 36 (7 days after second dose)
Percentage of participants with unsolicited adverse events occurring up to 28 days after last i.m. vaccination (phase 1a) | Up to Day 57 (28 days after second dose)
Percentage of participants with adverse events of special interest occurring up to last visit (phase 1a) | Up to Day 197 (196 days after first dose)
  Adverse events of special interest represent a subset of AEs that include autoimmune diseases and other systemic disorders of interest which could potentially have an autoimmune etiology
Percentage of participants with serious adverse events (SAEs) occurring up to last visit (phase 1a) | Up to Day 197 (196 days after first dose)
Percentage of participants with solicited adverse events occurring up to seven days after i.n. mucosal recall (phase 1a) | Day 85 up to Day 92 (7 days after mucosal recall)
  This outcome is only measured for phase 1a Arm 4a and Arm 4b. Solicited adverse events related to mucosal recall consist of local and systemic reactions
Percentage of participants with unsolicited adverse events occurring up to 28 days after i.n. mucosal recall (phase 1a) | Day 85 up to Day 113 (28 days after mucosal recall)
  This outcome is only measured for phase 1a Arm 4a and Arm 4b
Percentage of participants with solicited injection site reactions recorded up to seven days after each vaccination (i.m. or i.d.) (phase 1b) | Up to Day 8 (7 days after first dose) and Day 29 up to Day 36 (7 days after second dose)
Percentage of participants with solicited systemic reactions recorded up to seven days after each vaccination (i.m. or i.d.) (phase 1b) | Up to Day 8 (7 days after first dose) and Day 29 up to Day 36 (7 days after second dose)
Percentage of participants with unsolicited adverse events occurring up to 28 days after last vaccination (phase 1b) | Up to Day 57 (28 days after second dose)
Percentage of participants with adverse events of special interest occurring up to last visit (phase 1b) | Up to Day 281 (280 days after first dose)
  Adverse events of special interest represent a subset of AEs that include autoimmune diseases and other systemic disorders of interest which could potentially have an autoimmune etiology
Percentage of participants with SAEs occurring up to last visit (phase 1b) | Up to Day 281 (280 days after first dose)
Percentage of participants with solicited adverse events occurring up to seven days after i.n. mucosal recall (phase 1b) | Day 211 up to Day 218 (7 days after mucosal recall)
  Solicited adverse events related to mucosal recall consist of local and systemic reactions
Percentage of participants with unsolicited adverse events occurring up to 28 days after i.n. mucosal recall (phase 1b) | Day 211 up to Day 239 (28 days after mucosal recall)
Frequencies of H107e-specific CD4+ T-cells producing any combination of Th1 cytokines (IFN-γ, TNF, and/or IL-2) induced by H107e/CAF®10b vs. placebo and vs. H107e/CAF®10b + BCG before vaccination (Day 1) and 2 weeks after 2nd vaccination (phase 1b) | Day 1 and Day 43
  Whole blood ICS is used to evaluate this outcome

SECONDARY OUTCOMES:
Frequencies of H107e-specific IFN-γ producing T-cells before first i.m. vaccination and two weeks after the second i.m. vaccination (phase 1a) | Day 1 and Day 43
  ELISpot assay on PBMCs is used to evaluate this outcome
Frequencies of BCG-specific CD4+ T-cells producing any combination of Th1 cytokines (i.e., IFN-γ, TNF and/or IL-2) induced by H107e/CAF®10b + BCG vs. BCG alone (Day 1 and 43) (phase 1b) | Day 1 and Day 43
  Whole blood ICS is used to evaluate this outcome

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Churchyard, PhD, Study Chair — Aurum Institute; Rasmus Mortensen, PhD, Study Chair — Statens Serum Institut
Locations (1):
- Aurum Institute, Pretoria, Gauteng, South Africa